CLINICAL TRIAL: NCT06712446
Title: A Pilot Study of Transcranial Magnetic Stimulation Plus Episodic Future Thinking for Methamphetamine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Heather E. Webber, PhD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HSC-MS-24-0886
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Methamphetamine Use Disorder
Keywords: delay discounting; methamphetamine; brain stimulation; episodic future thinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- highfrequency rTMS+EFT (Experimental)
  Interventions: Behavioral: EFT; Device: high frequency rTMS
- sham rTMS+EFT (Sham Comparator)
  Interventions: Behavioral: EFT; Device: sham frequency rTMS

INTERVENTIONS:
Behavioral: EFT — Participants will identify three personalized and rewarding future events not related to drug use that take place 1 week, 1 month, and 6 months in the future. Participants will be asked to rate the vividness of each personalized future positive event on a 5-pt Likert scale.A brief and personalized EFT prompt will be created for each future event . Personalized EFT prompts will be presented during delay discounting and MA demand assessments following EFT training. Participants will also receive daily text/email messages with these prompts, reminding them to engage in EFT, vividly reexperience their future events, over the week following EFT training.
Device: high frequency rTMS — TMS will be delivered with a MagVenture Mag Pro R30 with the Cool-B70 A/P coil with active liquid cooling . For dlPFC, we will measure position F3. The first session will begin with the acquisition of the resting motor threshold on the contralateral hand. Intermittent theta burst stimulation (iTBS) (triplet 50 Hz bursts, repeated at 5 Hz, 2 sec on and 8 sec off; 600 pulses per session) will be delivered at 110% of the resting motor threshold (RMT) and will last ~3 minutes. Participants will receive 2 sessions of iTBS to the dlPFC brain region with a 15-20-minute interval between sessions
  Arms: highfrequency rTMS+EFT
Device: sham frequency rTMS — Participants will receive sham TMS to the dlPFC. They may feel the TMS from the A/P coil electrodes, but there will not be any real stimulation of the brain.
  Arms: sham rTMS+EFT

SUMMARY:
The purpose of this study is to assess impact of repetitive transcranial magnetic stimulation (rTMS)+Episodic Future Thinking (EFT) vs. sham rTMS+EFT on delay discounting and methamphetamine (MA) demand, on vividness of future positive events during EFT training and on frequency of episodic thinking during the week following EFT training

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for primary methamphetamine use disorder
* Be fluent in English and able to understand the consent form

Exclusion Criteria:

* Current DSM-5 diagnosis for any illicit substance use disorder other than methamphetamine and marijuana
* Current DSM-5 diagnosis of moderate or greater severity for alcohol and marijuana use disorder
* In the opinion of the PI, the presence of any medical, neurological, psychiatric (e.g., psychotic or bipolar disorder), or physical condition, disease, or illness that, may: (a) compromise, interfere, limit, effect or reduce the subject's ability to complete the study; or (b) adversely impact the safety of the subject or the integrity of the data
* Has current or recent (within 3 months of potential enrollment) suicidal ideation, suicidal behavior, homicidal ideation or a homicidal plan sufficient to raise subject safety concerns based on the following assessments according to the PI:

  1. Structured Clinical Interview for DSM-5 (SCID-5)
  2. Columbia-Suicide Severity Rating Scale (C-SSRS) Screening - Answers YES to Questions 3, 4, 5, or 6
  3. Assault & homicidal danger assessment tool - Key to danger >1
* Medical implants contraindicating TMS (i.e., aneurysm clips or coils, stents, implanted stimulators, implanted vagus nerve or deep brain stimulators, implanted electrical devices such as pacemakers or medication pumps, electrodes for monitoring brain activity, cochlear implants for hearing, any magnetic implants, bullet fragments, any other metal device or object implanted in your body closer than 30 cm from the coil)
* History of brain surgery
* History of an intracranial lesion or any medical or neurological diagnosis/condition associated with increased intracranial pressure (i.e., Idiopathic Intracranial Hypertension/Pseudotumor Cerebri) OR any of the following symptoms within 30 days of enrollment: headaches > 15 days/month, loss of vision or decreased vision
* Moderate-to-severe heart disease
* History of stroke
* Is taking any antidepressant or antipsychotic medication at a dose above the maximum recommended dose or at a dose deemed to be potentially unsafe according to the PI; has taken any of the following medications, which are known to increase the risk of seizures, within 1 week of study enrollment; or does not agree to abstain from taking the following medications during study participation:

  1. clozapine
  2. chlorpromazine
  3. bupropion
  4. clomipramine hydrochloride
  5. amoxapine
  6. maprotiline hydrochloride
  7. diphenhydramine
  8. stimulants other than methamphetamine including the following: Dextroamphetamine and amphetamine, Dextroamphetamine, Lisdexamfetamine dimesylate, Cocaine, Methylphenidate,
  9. tramadol
  10. isoniazid
* Personal history of epilepsy or seizure disorder and/or family history including a first-degree relative
* Serious head injury with loss of consciousness
* Impending incarceration
* Pregnant or nursing females
* Inability to read, write, or speak English
* For adolescent aged participants (18-21 only): any risk factor for neurocardiogenic syncope (history of syncope/presyncope related to noxious stimuli, anxiety, micturition, or posture)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of delay discounting as assessed by the 5-Trial adjusting Delay Discounting Task | before TMS+EFT, after TMS+EFT, 7-day follow-up
  This 5 item questionnaire measures the extent to which participants devalue a reward as the delay to its receipt increases.This task presents choices between $500 now vs. $1,000 after a delay.The discount rate k quantifies how rapidly the value of a delayed reward decreases with time.Low k Indicates patience or low impulsivity - greater willingness to wait for larger rewards.High k Indicates impatience or high impulsivity - preference for immediate rewards over delayed ones.
Change in MA Demand as assessed by the Drug Purchasing Task | before TMS+EFT, after TMS+EFT, 7-day follow-up
  MA demand will be assessed by asking participants how many grams of MA they would purchase to use over the course of a weekend (Friday night to Sunday night) as a function of increasing price ($0 to $10000) Demand is the maximum quantity of Methamphetamine consumed if the drug was free measured in grams or dollar amount
EFT Vividness as assessed by the Vividness Scale | measured during EFT training on study day 1
  This is a single item questionnaire and is scored on a 5-point Likert scale from 1(not vivid at all) to 5( extremely vivid) for a maximum score of 5, higher score indicating more vivid outcome
EFT Engagement as assessed by the Engagement Scale | 7-day follow-up
  This is a single item questionnaire and is scored on a 4-point Likert scale 1-4 asking how often each individual engaged in EFT (i.e., every day, most days, some days, no days), higher score indicating more engagement

SECONDARY OUTCOMES:
Change in prospective memory as assessed by the Prospective and Retrospective Memory Questionnaire (PRMQ) | before TMS+EFT, after TMS+EFT, 7-day follow-up
  This is a 16 item questionnaire and each is scored on a 5-point Likert scale from 1(never) to 5(very often) for a maximum score of 80, higher score indicating better outcome
Change in prospective memory (PM) as assessed by the behavioral PM task | before TMS+EFT, after TMS+EFT, 7-day follow-up
  The percentage of correct target identifications on the PM task
Number of days of Methamphetamine use as assessed by the time line follow back (TLFB) method | 7-day follow-up
Amount of Methamphetamine used in grams as assessed by the time line follow back (TLFB) method | 7-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heather Webber, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided